CLINICAL TRIAL: NCT02372890
Title: Validation of High-resolution PET/CT for the Pretherapeutic Lymphnode Staging of Head/Neck Cancer
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 277/2014
Record Dates: First submitted 2015-01-19; First posted 2015-02-26 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Otorhinolaryngeal Neoplasms; Cancer of Head and Neck
Keywords: Otorhinolaryngeal Neoplasms; Cancer of Head and Neck; Head and Neck Squamous Cell Carcinoma; Positron Emission Tomography; PET/CT; FDG
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Patients with head and neck squamous cell carcinoma with advanced primary tumor stages (cT3 or cT4), clinical suspicion of cervical lymph node metastases, cervical lymph node metastasis of unknown primary tumor (CUP) or patients with tumor recurrence scheduled for neck dissection.

SUMMARY:
In head and neck squamous cell carcinoma (HNSCC), the presence of lymph node metastases in addition to free resection margins following surgical resection of the primary tumor is an important prognostic factor, and may impact planning of surgery as well as of radiotherapy. Until now, imaging modalities including PET/CT and MRI did not allow to exclude especially small lymph node metastases.

Compared to standard whole-body PET/CT acquisition techniques, high-resolution (HR) head and neck PET/CT acquisitions promise improved detection of lymph node metastases in head and neck squamous cell carcinoma (HNSCC). This prospective study aims to determine the sensitivity and specificity of lymph node staging with HR FDG-PET/CT in HNSCC by correlating PET/CT with histopathology after neck dissection. HR PET/CT may have a relevant impact on the therapeutic concept, and the planning and dose prescription of radiotherapy.

DETAILED DESCRIPTION:
In head and neck squamous cell carcinoma (HNSCC), the presence of lymph node metastases in addition to free resection margins following surgical resection of the primary tumor is an important prognostic factor, and may impact planning of surgery as well as of radiotherapy. Neck dissection and histopathology are regarded as diagnostic standard procedures to define the lymph node status in patients with HNSCC. Occult lymph node metastases after imaging have been described in up to 46% of patients, e.g. in patients with cancer of the tongue.

Although neck dissection generally has a low rate of intra- and postoperative complications, a small but statistically significant group of patients suffers from surgery-related side effects such as lymphedema, chronic pain syndromes and injury of cranial nerves with paralysis (shoulder lift and mouth angle). Therefore it would be desirable to spare diagnostic neck dissection in patients without macroscopic lymph node metastasis. However, the sensitivity and/or specificity of the non-invasive imaging techniques available up to now, including positron emission tomography (PET) and magnetic resonance imaging (MRI), did not allow to exclude lymph node metastases, which is especially true for small metastases. Therefore, imaging is not able to replace the histological examination of the cervical lymph nodes and have limited impact on the therapeutic concept, the surgical planning and the planning and dose prescription of radiotherapy.

Acquisition techniques and image quality of PET (with the glucose analog F-18-fluorodeoxyglucose (FDG)) and the combined examination with computed tomography (PET/CT) were considerably improved with last generation PET/CT machines. New generation PET/CT machines provide significantly improved image quality and image resolution image, and probably higher sensitivity to detect smaller lesions. However, in the face of an expected increase of detected metabolically active cervical lymph nodes by high-resolution (HR) PET/CT, a diagnostic problem in terms of a potentially increased number of false-positive lymph nodes arises, e. g. due to an inflammatory lymphadenopathy.

Until now there are no evidence-based criteria to classify small metabolically active lymph nodes detected by HR PET/CT. Hence, a correlation of PET/CT findings and histopathology of cervical lymph metastases and inflammatory lymph nodes in patients with HNSCC is required to develop diagnostic criteria for HR PET/CT and to exploit the diagnostic potential of HR PET/CT.

Modern concepts of radiotherapy planning for neck lymph node metastases increasingly take into consideration the metabolic and morphological information of PET/CT for target volume definition. Detailed information on the diagnostic performance of HR PET / CT are of importance for the dose prescription of intensity-modulated radiotherapy (IMRT). In radiotherapy side effects depend significantly on the dose and the irradiation volume. Modern radiation techniques, especially IMRT, allow for highly-conformal radiation therapy with steep dose gradients to protect organs such as the salivary glands, and to reduce side effects of radiotherapy. On the other hand modern radiotherapy concepts carry the risk to fail due to non-inclusion of subclinical lymph node metastases in the target volume. HR PET/CT may allow to minimize out-of-field recurrences caused by incorrect target volume contouring or dose prescription. Evidence-based data on the diagnostic accuracy of HR PET/CT with special regard to small lymph node metastases are needed to clarify the potential role of HR PET/CT for radiation treatment planning.

Objective:

* To determine the sensitivity, specificity, accuracy, PPV and NPV of lymph node staging with HR PET/CT in patients with HNSCC
* To determine the sensitivity, specificity, accuracy, PPV and NPV of HR PET/CT for lymph node metastases of different size in patients with HNSCC
* To determine the detection rate of distant metastases by PET/CT in patients with HNSCC
* To develop diagnostic criteria for the multi-modal lymph node staging with HR PET/CT in patients with HNSCC
* To evaluate the potential impact of HR PET/CT on radiation treatment planning

Methods:

Patients with HNSCC are managed according to clinical recommendations of the interdisciplinary tumor board. Elective patients receive selective, modified radical or radical neck dissection of the relevant lymph node region according to clinical routine standards at the Inselspital Bern. The neck dissection must be carried out within a maximum of 6 weeks after the PET / CT examination.

As part of the neck dissection the lymph nodes will be sent to the Institute of Pathology separated by level and side by topographic markers (cranial / caudal, medial / lateral). The histological examination of the removed lymph nodes serves as reference standard for the analysis of PET/CT image data, and calculation of the diagnostic accuracy of HR PET/CT.

Theoretical radiation treatment plans are generated based on conventional imaging, whole-body PET/CT and HR PET/CT protocols to determine the impact of PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck squamous cell carcinoma (HNSCC), fulfilling one or more of the following criteria:

  * Advanced primary tumor stage (cT3 or cT4)
  * Clinical suspicion of neck lymph node metastases
  * Cervical lymph node metastases of unknown primary tumor (CUP)
  * Tumor recurrence
* Mature adult
* Written informed consent

Exclusion Criteria:

* Inoperability
* Histologically verified cervical lymph node metastases of other tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck squamous cell carcinoma undergoing routine PET/CT staging or restaging and sheduled for neck dissection according to the decision of the interdisziplinary tumor board.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2012-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy (sensitivity, specificity, accuracy, NPV und PPV) of HR PET/CT in comparison to the histopathological reference standard | At baseline

SECONDARY OUTCOMES:
Diagnostic accuracy (sensitivity, specificity, accuracy, NPV und PPV) of PET/CT according to the size of lymph node metastases | At baseline
Number of patients where PET/CT results in a change of gross tumor volume (GTV) and/or dose prescription | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Arnold, Prof. Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Dept. of Nuclear Medicine, Bern University Hospital, Bern, Bern, Switzerland